CLINICAL TRIAL: NCT02274181
Title: An Open-Label, Single-Dose Study to Assess the Absorption, Metabolism, Excretion, and Mass Balance of Radiolabeled Androxal in Healthy Male Subjects After Oral Administration
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Repros Therapeutics Inc. (Industry)
Collaborators: Celerion (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZA-112
Record Dates: First submitted 2014-10-06; First posted 2014-10-24 (Estimated); Last update posted 2015-03-12 (Estimated); Status verified 2015-03

CONDITIONS: Secondary Hypogonadism
MeSH Terms: conditions — Hypogonadism | interventions — Enclomiphene

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 25 mg (approximately equivalent to [(~]) 500 nanocurie (Experimental): A single 25 mg (approximately equivalent to [(~]) 500 nanocurie [nCi]) dose of [14C]Androxal
  Interventions: Drug: Androxal

INTERVENTIONS:
Drug: Androxal

SUMMARY:
The purpose of this study is to investigate the route(s) of elimination and mass balance of enclomiphene after oral administration of a single 25 mg (approximately equivalent to [(~]) 500 nanocurie [nCi]) dose of [14C]Androxal in healthy adult male subjects.

DETAILED DESCRIPTION:
The purpose of this study is to investigate the route(s) of elimination and mass balance of enclomiphene after oral administration of a single 25 mg (approximately equivalent to [(~]) 500 nanocurie [nCi]) dose of [14C]Androxal in healthy adult male subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy, adult, male subjects, 19 60 years of age, inclusive, at screening
2. Continuous non smoker who has not used nicotine containing products for at least 3 months prior to dosing
3. Body mass index (BMI) ≥ 25.0 and ≤ 42.0 kg/m2 at screening
4. Medically healthy with no clinically significant medical history, physical examination, laboratory profiles, vital signs or ECGs, as deemed by the PI
5. A non vasectomized, male subject must agree to use a condom with spermicide or abstain from sexual intercourse during the study until 90 days beyond the last dose of study drug. (No restrictions are required for a vasectomized male provided his vasectomy has been performed 4 months or more prior to study start. A male who has been vasectomized less than 4 months prior to study start must follow the same restrictions as a non vasectomized male)
6. Must agree not to donate sperm from dosing until 90 days after dosing
7. Understands the study procedures in the informed consent form (ICF), and be willing and able to comply with the protocol

Exclusion Criteria:

1. Subject is mentally or legally incapacitated or has significant emotional problems at the time of the screening visit or expected during the conduct of the study
2. History or presence of clinically significant medical or psychiatric condition or disease in the opinion of the PI
3. History of any illness that, in the opinion of the PI, might confound the results of the study or poses an additional risk to the subject by their participation in the study
4. History or presence of alcoholism or drug abuse within the past 2 years prior to screening
5. History or presence of hypersensitivity or idiosyncratic reaction to the study drug or related compounds (e.g., clomiphene citrate)
6. History or presence of:

   * Renal disease or a history of renal dysfunction;
   * Liver disease or a history of liver dysfunction;
   * Uncontrolled thyroid or adrenal dysfunction or in the presence of an organic intracranial lesion such as a pituitary tumor;
   * Previous history of deep vein thrombosis, pulmonary embolism or a high risk for stroke
   * Conditions which are known to be exacerbated by testosterone replacement or are driven by androgen sensitivity
7. Regularly have less than 1 bowel movement every 2 days
8. Recent history (within 2 weeks of Day -1) of abnormal bowel habits, such as diarrhea, loose stools, or constipation
9. Positive urine drug or alcohol results at screening or check in
10. Positive urine cotinine at screening
11. Positive results at screening for HIV, HBsAg or HCV
12. Poor metabolizer for CYP2D6 based on genotyping for CYP2D6 at screening (since CYP2D6 is key enzyme for enclomiphene drug metabolism).2
13. Unable to refrain from or anticipates the use of:

    * Any drug, including prescription and non prescription medications (including any drugs known to be significant inhibitors of CYP enzymes and/or P gp and/or OATP), herbal remedies, or vitamin supplements beginning 14 days prior to dosing of study drug and throughout the study. Acetaminophen (up to 2 g per 24 hour period) and Milk of Magnesia (≤ 60 mL per day) may be permitted during the study
    * Any drugs known to be significant inducers of CYP enzymes and/or P gp, including St. John's Wort, for 28 days prior to dosing of study drug and throughout the study. Appropriate sources will be consulted by the PI or designee to confirm lack of PK/pharmacodynamics (PD) interaction with study drug
14. Have been on a diet incompatible with the on study diet, in the opinion of the PI, within the 28 days prior to dosing of study drug, and throughout the study
15. Have received radiolabeled substances or have been exposed to radiation sources over the past 12 months or is likely to receive radiation exposure or radioisotopes within the next 12 months such that participation in this study would increase their total exposure beyond the recommended levels considered safe (i.e., weighted annual limit recommended by the ICRP of 3000 mrem)
16. Donation of blood or significant blood loss within 56 days prior to dosing of study drug
17. Plasma donation within 7 days prior to dosing of study drug
18. Participation in another clinical trial within 28 days prior to dosing of study drug. The 28 day window will be derived from the date of the last blood collection or dosing, whichever is later, in the previous study to Day 1 of the current study

Ages: 19 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2014-12; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Percentage of Androxal excreted via the urine, feces and blood | 8 Days
  Determined by AMS lab by analysis of all excreted samples

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Cook, MD, Principal Investigator — Celerion
Locations (1):
- Celerion, Lincoln, Nebraska, United States